CLINICAL TRIAL: NCT05259774
Title: A Multicenter, Double Blind, Randomized, Vehiclecontrolled Clinical Study Evaluate the Efficacy and Safety of Relizema Cream in the Management of Atopic Dermatitis in Paediatric Patients.
Brief Title: Clinical Investigation on the Efficacy and Safety of Relizema Cream in Paedriatric Patients
Acronym: YOUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReGl/21/Rcr-Dpe/001
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: cream; paediatric patients
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: multicenter, double blind, controlled versus placebo, pre-market clinical followup investigation
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly allocated to one of the following treatment groups: Relizema cream and vehicle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relizema cream (Experimental): Relizema cream, topically applied twice a day in all the affected areas for three cycles of 13 (±2) consecutive days.
  Interventions: Device: Relizema cram
- Vehicle (No Intervention): Cream, topically applied twice a day in all the affected areas for three cycles of 13 (±2) consecutive days.

INTERVENTIONS:
Device: Relizema cram — Relizema cream is a CE marked, Class IIa medical device, dermatological cream for topical use indicated for symptomatic treatment of dermatitis and erythema. Relizema cream is indicated for the treatment of itching and flushing associated with different types of dermatitis, including atopic dermatitis.
  Arms: Relizema cream

SUMMARY:
The scope of this multicenter, double blind, randomized, vehicle-controlled clinical investigation is to evaluate and confirm the performance and safety of the Relizema cream in the improvement of the dermatitis severity in paediatric patients. The disease severity will be clinically measured through the Investigator Global Assessment (IGA) after 42 days of treatment.

DETAILED DESCRIPTION:
This is a Pre Market Study to evaluate and confirm the performance of the RelizemaTM cream in the improvement of the dermatitis severity, assessed through a clinical parameter, the Investigator's Global Assessment (IGA) at baseline and at Visit 3, compared to vehicle.

To evaluate the performance of the RelizemaTM cream, compared to placebo in the eczema improvement through the EASI.

The safety objectives is to evaluate the local and general tolerability of Relizema cream compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Release of the written informed consent obtained prior to any study-related procedures, by both the parents/the guardian;
* Male and female infants, children, adolescent aged between 6 months and 16 years, inclusive;
* Presence of atopic dermatitis (AD) of mild-moderate severity:
* IGA score 2 (=mild) or
* IGA score 3 (=moderate)
* Patients with a baseline score for itch at least 4 on the NRS
* Patients/parents/guardian able to comprehend the full nature and the purpose of the investigation, and able to comply with the requirements of the entire investigation (including ability to attend the planned visits according to the time limits), based on Investigator's judgement

Exclusion Criteria:

* Severe dermatitis at inclusion;
* Pregnant and breastfeeding patients;
* Concomitant other skin disorders including skin infections;
* Use of antibiotics in the past 7 days;
* History of congenital or acquired immunodepression;
* Immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, any typology of lupus, rheumatoid arthritis) which could place the patient at risk or interfere with study results;
* Use of any topic or systemic drug for dermatitis in the past 10 days;
* Use of any topic emollient product for dermatitis in the 2 days before study treatment start;
* Any systemic treatment or procedure that could influence dermatitis activity within the past 30 days (or 5 half-lives);
* Use of any corticosteroids, immunosuppressant drugs or immunotherapy within the past 30 days (or 5 half-lives);
* Use of oral antihistamines and antidepressants in the past 30 days;
* Patients with any other clinically significant or unstable concurrent disease or skin condition or general condition that, in the Investigator's opinion, might interfere with the study evaluations;
* Allergy, sensitivity or intolerance to the components of the investigational device formulations ingredients;
* Concomitant or previous participation in other interventional clinical study in the past 3 months;
* Patients planning sun exposure or tanning booths or UV sources throughout the course of the study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Stingeni, Principal Investigator — Santa Maria della Misericordia Hospital
Locations (1):
- Luca Stingeni, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relizema Cream | Vehicle
Started | 25 | 25
Completed | 24 | 23
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients were divided into 3 groups: infants from 6 months to 2 years, children from 3 to 11 years and adolescents from 12 to 16 years inclusive.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relizema Cream | Vehicle | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.33 (4.97) | 6.42 (4.45) | 6.38 (4.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 15 | 16 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  Italy | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate and Confirm the Performance of the Relizema Cream in the Improvement of the Dermatitis Severity in Paediatric Patients.
Description: The disease severity will be clinically measured through the Investigator Global Assessment (IGA) for dermatitis after 28 days of treatment, compared to vehicle.
Time Frame: 28 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
Participants | 17 | 13

2. Secondary Outcome: To Evaluate the Performance of the Relizema Cream, Compared to Placebo,
Description: To evaluate the performance of the Relizema cream, compared to placebo, in the improvement of dermatitis severity (IGA) after 14 and 42 days of treatment
Time Frame: after 14 and 42 days of treatment, 42 days reported
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
Participants | 12 | 10

3. Secondary Outcome: To Evaluate the Eczema Improvement
Description: To evaluate the eczema improvement through the EASI (Eczema Area and Severity Index) score
Time Frame: after 14, 28 and 42 days of treatment, reported after 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
Participants | 18 | 14

4. Secondary Outcome: To Evaluate the Media in Itching, Burning, Pain and Pruritus at Visits
Description: To evaluate itching as reported by the patient at visits by the Numerical Rating Scale (NRS that is a numeric scale from 0 to 10, 0 is the best result, 10 is the worst), in the two treatment groups
Time Frame: after 14, 28 and 42 days of treatment, day 42 reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
units on a scale | 5.45 (6.62) | 4.31 (6.26)

5. Secondary Outcome: To Evaluate Improvement in the Quality of Life (QoL) of the Subject Related to His/Her Dermatitis
Description: To evaluate the QoL improvement of the patient related to his/her dermatitis, through the Children Dermatology Life Quality Index (CDLQI) questionnaire in the two treatment groups; The questionnaire asks for 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week.
  Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
  Global score:
  0-1 = No effect on patient's life 2-5 = Small effect 6-10 = Moderate effect 11-20 = Very large effect 21-30 = Extremely large effect. The CDQLI was compiled by the patient at each visit. Young children were supported for the questionnaire compilation by the parents/guardian, if necessary)
Time Frame: after 14, 28 and 42 days of treatment, reported 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
units on a scale | 2.42 (1.67) | 1.83 (1.86)

6. Secondary Outcome: To Evaluate the Patient's Adherence to Treatment
Description: Units on a scale of partecipants with an improvement in the dermatitis severity
Time Frame: 42 days
Population: Treatment adherence was assessed by counting the applications reported in the patient's diary and dividing by the total number of applications. The percentage of applications applied is reported
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
percentage of adherence | 97.46 (5.13) | 96.96 (7.32)

7. Secondary Outcome: To Evaluate the Need of a Rescue Treatment (as Indicated by the Investigator) to Manage AD Flare;
Description: To evaluate the need of a rescue treatment (as indicated by the Investigator) to manage AD flare;
Time Frame: 42 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
Participants | 21 | 16

8. Secondary Outcome: To Evaluate the Patient's Global Evaluation of Performance of Relizema Cream, Compared to Placebo
Description: To evaluate the patient's global evaluation on performance of the study product performed by means of a 7-items scale (where 1 = very much improved, 2 = improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = worse, 7 = very much worse)
Time Frame: at the end of the study ( day 42)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relizema Cream | Vehicle
Number analyzed (Participants) | 25 | 25
units on a scale | 5.29 (4.73) | 3.53 (4)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Relizema Cream | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT05259774/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT05259774/ICF_001.pdf